CLINICAL TRIAL: NCT00691834
Title: ReNEW: A Phase 2, Randomized, Placebo-Controlled, Double-Blinded Study of the Efficacy and Safety of Autologous Bone Marrow Mononuclear Cell Transfer for Myocardial Salvage in Acute Myocardial Infarction
Brief Title: Safety and Efficacy on Cell-based Therapy in Patients With Recent Large Acute Myocardial Infarction
Acronym: ReNeW
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never received IRB approval. Study was never pursued.
Sponsor: Duke University (Other)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00003467
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2012-11

CONDITIONS: Acute Myocardial Infarction; Heart Failure
Keywords: Magnetic resonance Imaging
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intracoronary delivery of unfractionated bone marrow mononuclear cells
  Interventions: Biological: Intracoronary delivery of unfractionated bone marrow mononuclear cells
- 2 (Placebo Comparator): Intracoronary delivery of placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Intracoronary delivery of unfractionated bone marrow mononuclear cells — Maximal intracoronary cell dose: 50 x 10e7 cells diluted in 10 ml Maximal intracoronary volume: 10 ml (diluted in plasma and culture medium)
  Arms: 1
Biological: Placebo — Plasma and culture medium (10 ml)
  Arms: 2

SUMMARY:
The purpose of this study is to test bone marrow mononuclear cells for patients with recent heart attack who are at high risk of experiencing heart failure. This study drug is made of you own cells. Studies similar to this one have suggested that the use of cell-based transfer after heart attack can improve the recuperation of the heart. The purpose of this study is to assess whether cell transfer can improve the healing of the heart after a heart attack.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age and no more than 80 years of age.
* Acute ST-segment elevation MI
* Symptoms suggestive of acute MI
* ≥ 2mm ST-segment elevation in 2 or more precordial leads or ≥ 1mm in or more limb leads or new left bundle branch block
* Time from symptom onset to enrollment < 120 hours
* Left ventricular dysfunction by contrast ventriculography or echocardiography
* EF above 25 % and lower than 40%
* Focal wall motion akinesis or dyskinesis
* Clearly identifiable infarct artery
* Patent infarct artery (TIMI flow grade 2 or 3) of ≥ 2 mm in diameter following successful stent placement

Exclusion Criteria:

* Planned treatment with bypass surgery or prior CABG
* Multi-vessel PCI
* Prior myocardial infarction by history or presence of pathologic Q-waves
* Active cardiogenic shock: mechanical ventilation, IABP, or vasopressors/inotropes
* Successful reperfusion < 3 hrs from symptom onset
* Prior MI or significant chronic heart failure
* Pacemaker/defibrillator
* Contraindication to MRI (metallic foreign body, claustrophobia, inability to lie flat)
* Significant hepatic dysfunction or renal insufficiency (estimated creatinine clearance<25 and/or serum Cr >2.5 mg/dl)
* Baseline hematocrit < 30
* Pregnancy, or lactation/parturition within the past 30 days
* Active or planned treatment with chemotherapy
* Anticipated difficulty with 90-day follow-up
* Evidence of a serious, active infection in the opinion of the investigator including, but not limited to subjects who are HIV, hepatitis B or C positive
* Any known severe hematological disease, malignancy, systemic or life threatening disorder that would be incompatible with the trial
* Previous enrollment in this trial
* Participation in an investigational drug or device study within the past 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Difference in the change of left ventricular ejection fraction between placebo-treated and cell-treated patients | baseline and 90 days
Occurence of arrhythmia, heart failure and death | 1 year

SECONDARY OUTCOMES:
Improvement in regional left ventricular function | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Christopher B Granger, MD, Principal Investigator — Duke Clinical Research Institute; Marc E Jolicoeur, MD MSc, Principal Investigator — Duke Clinical Research Institute